CLINICAL TRIAL: NCT04169958
Title: Suicide Risk Assessment by Digital Means
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Nadav Goldental, Principal Investigator, The Chaim Sheba Medical Center
Other Study IDs: SHEBA-18-5152-NG-CTIL
Record Dates: First submitted 2018-12-22; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: safe mood — A tablet application that developed for this study. In addition, sensors are used to examine the possibility of using the system to assess the risk of suicide

SUMMARY:
This study is an observational study, without intervention. Using a tablet application that developed for this study. In addition, sensors are used to examine the possibility of using the system to assess the risk of suicide. It should be noted that this is a pilot study, only for a wider study involving a larger number of patients.

The system developed for the benefit of this study is based on a smartphone application installed on a standard Smartphone device that will be found in the ED or by the examiner. The system collects data from five channels one by one (the information collected from each channel is collected separately).

The data recorded from the various channels is saved on the tablet device. Then, the information transferred to the database using a cable. A statistical analysis of the data from the various channels is carried out in order to assess suicidal behavior.

After the statistical analysis, correlations will be examining between the results of the measurements and the results of the accepted questionnaires for the assessment of suicidality, which will be performed simultaneously.

Note that the duration of participation is the duration of the measurements, ie a single session that lasts up to two hours The duration of the participants in the study is determined by the time of the measurements, ie a single session lasting up to two hours.

ELIGIBILITY:
Inclusion Criteria:

* Every patient who is examined in the psychiatric ward at the Sheba Medical Center
* Proper ability to give informed consent

Exclusion Criteria:

* A patient who is not independent and without an active therapist / guardian involved in the treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit a total sample of N=50 in three stages:
  * Males and Females
  * 30 patients aged 12 - 18 years old (20% of the study sample) Participants will be recruited from the psychiatric ER (~50%), outpatient clinics (~20%), and inpatient wards (~30%) at the Sheba Medical Center, the largest hospital in Israel, serving a very large, demographically heterogenic and socioeconomically diverse population.
  * Psychiatric diagnosis: None, Affective Disorder, PTSD, ADHD, Personality Disorder, Anxiety Disorder, OCD.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-11-29 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlations between collected digital data and suicidality rating score | 1.5 years
  Correlations between collected digital data and suicidality rating score.

IPD SHARING:
Plan to Share IPD: Undecided